CLINICAL TRIAL: NCT05362422
Title: Paired Associative Stimulation for Post- Spinal Cord Injury Neuropathic Pain
Brief Title: PAS for Post-SCI Neuropathic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Anastasia Shulga, Head of Department, Helsinki University Central Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TYH2020244
Record Dates: First submitted 2022-04-22; First posted 2022-05-05 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Spinal Cord Injury Cervical; Neuropathic Pain
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PAS (Experimental)
  Interventions: Device: long-term paired associative stimulation
- SHAM (Sham Comparator)
  Interventions: Device: sham long-term paired associative stimulation

INTERVENTIONS:
Device: long-term paired associative stimulation — Paired associative stimulation (PAS) administered 3-5 times per week for 4 weeks to upper limbs. PAS comprises transcranial magnetic stimulation (eXimia magnetic stimulator, Nexstim Ltd, Helsinki, Finland) and peripheral nerve stimulation (given with Dantec Keypoint® electroneuromyography device (Natus Medical Incorporated, Pleasanton, CA, USA)).
  Arms: PAS
Device: sham long-term paired associative stimulation — Sham transcranial magnetic stimulation and sham peripheral nerve stimulation.
  Arms: SHAM

SUMMARY:
The investigators have shown in incomplete SCI patients that long-term paired associative stimulation is capable of restoring voluntary control over some paralyzed muscles and enhancing motor output in the weak muscles. In this study, the investigators will administer long-term paired associative stimulation to patients with incomplete cervical level SCI and SCI- associated neuropathic pain, and investigate its effectiveness for neuropathic pain treatment.

ELIGIBILITY:
Inclusion Criteria:

* incomplete cervical spinal cord injury
* time from injury at least 1.5 years
* chronic SCI- induced neuropathic pain in the upper limb

Exclusion Criteria:

* Diagnosed brain damage, visible in MRI or CT.
* No activity in hands/fingers and no MEPs recorded from distal hand muscles.
* Epilepsy
* Metal inclusion in the head area
* High intracranial pressure
* Pacemaker
* Implanted hearing device
* Progressive diseases of spinal cord or brain (e.g. malignant tumors, degenerative diseases).
* Previous head or spinal cord injury affecting the motor performance of upper extremities.
* Congenital anomaly in the anatomical structure of spinal canal/cord or dura.
* Significant systemic disease or other condition that could cause neurological deficit, or may affect subject's capability to undergo investigation-related procedures.
* Acute severe infection.
* Contraindications for MRI.
* Current severe psychiatric diseases.
* Current chronic drug and/or alcohol abuse.
* Pregnancy.
* Pressure ulcer affecting the subject's capability to undergo the procedure safely

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2023-09-22 (Actual)

PRIMARY OUTCOMES:
Brief Pain Inventory | Change from baseline at 1 day after the intervention
  0-10 scale, 0 - no pain, 10 - worst possible pain.
Brief Pain Inventory | Change from baseline at 8 weeks after the intervention
  0-10 scale, 0 - no pain, 10 - worst possible pain.
Numeric Rating Scale | Change from baseline at 1 day after the intervention
  0-10 scale, 0 - no pain, 10 - worst possible pain.
Numeric Rating Scale | Change from baseline at 8 weeks after the intervention
  0-10 scale, 0 - no pain, 10 - worst possible pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Helsinki University Hospital, Helsinki, Finland

REFERENCES:
- [Background] Shulga A, Lioumis P, Kirveskari E, Savolainen S, Makela JP. A novel paired associative stimulation protocol with a high-frequency peripheral component: A review on results in spinal cord injury rehabilitation. Eur J Neurosci. 2021 May;53(9):3242-3257. doi: 10.1111/ejn.15191. Epub 2021 Mar 29. PMID 33738876
- [Background] Vaalto S, Nyman AL, Shulga A. Analgesic effect of paired associative stimulation in a tetraplegic patient with severe drug-resistant neuropathic pain: a case report. Scand J Pain. 2021 May 21;21(4):831-838. doi: 10.1515/sjpain-2021-0012. Print 2021 Oct 26. PMID 34019752